CLINICAL TRIAL: NCT00287742
Title: Double-blind, Placebo-controlled Clinical Trial of JK6476 (Risperidone) in Patients With Hallucinations and Delusions Associated With Alzheimer's Disease
Brief Title: A Study of the Effectiveness and Safety of Risperidone Versus Placebo in the Treatment of Patients With Hallucinations and Delusions Associated With Alzheimer's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: A decision was made to discontinue the study due to a change in the strategic direction of the company.
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003172
Record Dates: First submitted 2006-02-03; First posted 2006-02-07 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2010-11

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: risperidone; antipsychotic agents; Alzheimer's disease; dementia; psychosis
MeSH Terms: conditions — Alzheimer Disease; Dementia; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of risperidone (an antipsychotic medication) versus placebo for the treatment of patients with hallucinations and delusions associated with Alzheimer's disease.

DETAILED DESCRIPTION:
Dementia is frequently observed in the elderly, often associated with psychotic symptoms such as delusion or hallucination, or with behavioral disturbances such as aggressive behavior, wandering, and aimless behavior induced by the psychotic symptoms. Based on the results of preliminary clinical studies, risperidone can be expected to be beneficial for the treatment of psychotic symptoms and behavioral disturbances associated with Alzheimer's disease. This is a multicenter, randomized, double-blind, placebo-controlled study of risperidone tablets or placebo tablets taken twice daily over 9 weeks by patients with hallucinations and delusions associated with Alzheimer's disease. During the one week run-in period, patients take one tablet twice daily. During the 8 week double-blind period, the dose is given twice daily in a flexible dose regimen of 0.5 to 2 mg of risperidone per day, or placebo. The primary measure of effectiveness is the change in Behavioral Pathology in Alzheimer's Disease (BEHAVE-AD) psychotic symptom cluster score from baseline and intermediate visits to study end (Week 9) compared with placebo. BEHAVE-AD is a scale used for global assessment of symptoms associated with dementia. Additional assessments of effectiveness include the Cohen-Mansfield Agitation Inventory (CMAI), an assessment of aggressiveness and non-aggressiveness, and the Clinical Global Impression - Change (CGI-C), a measure of an improved or aggravated condition. Safety evaluations include the incidence of adverse events, physical examinations, electrocardiograms (ECGs), laboratory tests (biochemistry, hematology, and urinalysis), and assessment of extrapyramidal symptoms. The study hypothesis is that treatment twice daily with risperidone is more effective than placebo on measures of the BEHAVE-AD psychotic symptom cluster score in patients with hallucinations and delusions associated with Alzheimer's disease. Oral risperidone tablets 0.25 mg or placebo tablets twice daily, increasing in weekly increments of 0.5 mg/day to a maximum of 2 mg/day; total daily dosage will be maintained for 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's disease according to criteria of Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV)
* Mini-Mental State Examination (MMSE) score of not greater than 23
* Behavioral Pathology in Alzheimer's Disease (BEHAVE-AD) psychotic score of >=2 for any item in the psychotic cluster
* occurrence of hallucination or delusion after onset of symptoms of dementia at least 28 days before screening.

Exclusion Criteria:

* Patients with a disease that could significantly diminish cognitive function (e.g., Parkinsonism, Huntington's disease, Creutzfeldt-Jacob disease, dementia of Levy body type, vitamin B12 or folic acid deficiency)
* persistent dementia or amnestic disorders according to DSM-IV criteria
* occurrence of hallucination or delusion only while delirium is observed
* psychiatric symptoms induced by psychosis (e.g., schizophrenia, schizoaffective disorders, delusional disorders, depression or bipolar disorders)
* history of neuroleptic malignant syndrome (a rare psychotropic-drug reaction, which may be characterized by confusion, reduced consciousness, high fever or pronounced muscle stiffness)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2002-03; Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Change in Behavioral Pathology in Alzheimer's Disease (BEHAVE-AD) psychotic symptom cluster score from baseline and intermediate visits to study end (Week 9) compared with placebo.

SECONDARY OUTCOMES:
Changes in BEHAVE-AD total, subscales and items scores, changes in CMAI aggressiveness and non-aggressiveness item scores and changes in CGI-C from baseline and intermediate visits to study end (Week 9) compared with placebo. Safety evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.

REFERENCES:
- See also: A study of the effectiveness and safety of risperidone in the treatment of patients with hallucinations and delusions associated with Alzheimer's disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1082&filename=CR003172_CSR.pdf